CLINICAL TRIAL: NCT00198640
Title: Antimicrobial Resistance of Streptococcus Pneumoniae Carriage Strains Among Bangladeshi Neonates: Epidemiology, Determinants and Risk Factors
Brief Title: AMR of Streptococcus Pneumoniae Carriage Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: H.22.02.06.06.A1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-08

CONDITIONS: Infection
Keywords: animal antibiotics; human antibiotics
MeSH Terms: conditions — Infections

INTERVENTIONS:
Procedure: Antibiotic use

SUMMARY:
This study looks at the usage of human antibiotics for treatment of animals in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Bangladesh location

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mathuram Santosham, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health